CLINICAL TRIAL: NCT03731741
Title: Effect of Pentoxifylline Administration on Hemoglobin Level of Hemodialysis Patients
Brief Title: Does Oral Pentoxifylline Administration Improve Hemoglobin in Hemodialysis Patients?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sarah Abdel Mageed, Assistant lecturer of internal medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pentoxifylline in inflammation
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Anemia of Chronic Kidney Disease
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Group I: 29 patients (25 completed the study) that received the study agent (400mg of oral pentoxifylline daily for 6 months.), besides the appropriate weight-based dose of ESA (60-150I.U/kg/wk).
  Interventions: Drug: Pentoxifylline
- control group (No Intervention): Group II: 28 patients (25 completed the study) who did not receive pentoxifylline but they received the appropriate dose of ESA. They were used as a control group and compared to group1 concerning the primary and the secondary outcomes.

INTERVENTIONS:
Drug: Pentoxifylline — a known drug of xanthine derivatives used in intermittent claudication
  Other Names: Trental
  Arms: treatment group

SUMMARY:
Our study investigated the effect of using a known drug used in intermittent claudication (named pentoxifylline) as an adjuvant to erythropoietin stimulating agents to improve anemia of hemodialysis patients.

DETAILED DESCRIPTION:
Fifty out of 57 hemodialysis anemic patients were finally included. They were assigned to two groups of equal numbers. Oral Pentoxifylline 400mg once daily was added to the treatment group which was compared to the control group over a six months period regarding hemoglobin, hematocrit, serum albumin and CRP.

Inclusion criteria: (Patients with ESRD on HD who have hemoglobin <11 g/dl, taking Erythropoietin alfa 4000 -12000 I.U/wk and having a urea reduction ratio >65%.). There were 57 patients who met the inclusion criteria out of 158 patients.

Exclusion criteria: Iron deficiency anemia with transferrin saturation <30%, intact PTH>300pg/ml, vitamin B12 or folate deficiency (evidenced by macrocytosis), history of intolerance to pentoxifylline or other xanthine derivatives, recent retinal or cerebral hemorrhage or active peptic ulcer disease, pregnancy or breastfeeding, presence of systemic hematological disease or known hemoglobinopathy, major surgery, infection, acute myocardial infarction, or malignancy within the last three months and patients who refused to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* (Patients with ESRD on HD who have hemoglobin <11 g/dl, taking Erythropoietin alfa 4000 -12000 I.U/wk and having a urea reduction ratio >65%.). There were 57 patients who met the inclusion criteria out of 158 patients

Exclusion Criteria:

* Iron deficiency anemia with transferrin saturation <30%, intact PTH>300pg/ml, vitamin B12 or folate deficiency (evidenced by macrocytosis), history of intolerance to pentoxifylline or other xanthine derivatives, recent retinal or cerebral hemorrhage or active peptic ulcer disease, pregnancy or breastfeeding, presence of systemic hematological disease or known hemoglobinopathy, major surgery, infection, acute myocardial infarction, or malignancy within the last three months and patients who refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
hemoglobin difference | after 6 months from the start
  the difference in haemoglobin concentration between the pentoxifylline and control group at the end of the 6 months study period.

SECONDARY OUTCOMES:
difference in inflammatory markers | after 6 months from the start
  Difference in CRP and albumin levels between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Atef Taha, M.D, Study Director — Tanta university hospital
Locations (1):
- Tanta university hospital, Tanta, Egypt

REFERENCES:
- [Background] Del Vecchio L, Locatelli F. Anemia in chronic kidney disease patients: treatment recommendations and emerging therapies. Expert Rev Hematol. 2014 Aug;7(4):495-506. doi: 10.1586/17474086.2014.941349. PMID 25025373
- [Background] Kuragano T, Kitamura K, Matsumura O, Matsuda A, Hara T, Kiyomoto H, Murata T, Fujimoto S, Hase H, Joki N, Fukatsu A, Inoue T, Itakura Y, Nakanishi T. ESA Hyporesponsiveness Is Associated with Adverse Events in Maintenance Hemodialysis (MHD) Patients, But Not with Iron Storage. PLoS One. 2016 Mar 2;11(3):e0147328. doi: 10.1371/journal.pone.0147328. eCollection 2016. PMID 26933949
- [Background] Cooper A, Mikhail A, Lethbridge MW, Kemeny DM, Macdougall IC. Pentoxifylline improves hemoglobin levels in patients with erythropoietin-resistant anemia in renal failure. J Am Soc Nephrol. 2004 Jul;15(7):1877-82. doi: 10.1097/01.asn.0000131523.17045.56. PMID 15213276
- [Background] Gonzalez-Espinoza L, Rojas-Campos E, Medina-Perez M, Pena-Quintero P, Gomez-Navarro B, Cueto-Manzano AM. Pentoxifylline decreases serum levels of tumor necrosis factor alpha, interleukin 6 and C-reactive protein in hemodialysis patients: results of a randomized double-blind, controlled clinical trial. Nephrol Dial Transplant. 2012 May;27(5):2023-8. doi: 10.1093/ndt/gfr579. Epub 2011 Oct 3. PMID 21968012